CLINICAL TRIAL: NCT02902172
Title: NSAID Use in Postpartum Hypertensive Women
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit necessary number of patients
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Jennifer Goldkamp, MD, MD, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 26976
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Results first posted 2018-10-31 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Acetaminophen; Anti-Inflammatory Agents, Non-Steroidal; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen (Other): Patients will be monitored for change in blood pressure
  Interventions: Drug: Acetaminophen
- NSAID (Other): Patients will be monitored during their postpartum stay (typical 2 days) and then again at 1 week and 6 weeks (standard practice of care) with blood pressure measurements
  Interventions: Drug: NSAID

INTERVENTIONS:
Drug: Acetaminophen — Blood pressure will be monitored during postpartum stay (typical 2 days) and then again at 1 week and 6 weeks (standard practice of care) with blood pressure measurements
  Other Names: Tylenol
  Arms: Acetaminophen
Drug: NSAID — Blood pressure will be monitored during postpartum stay (typical 2 days) and then again at 1 week and 6 weeks (standard practice of care) with blood pressure measurements
  Other Names: Ibuprofen
  Arms: NSAID

SUMMARY:
Women who have the diagnosis of hypertension (pre-pregnancy and pregnancy induced) and deliver an infant via vaginal delivery will be placed into two groups in the postpartum period. One group will receive Ibuprofen for pain control and the other group will be given Tylenol. Blood pressures during the postpartum period will then be collected and compared in order to see if NSAIDs use increases blood pressure.

DETAILED DESCRIPTION:
The patients who have a vaginal delivery and have the diagnosis of hypertension in pregnancy will be randomized to either Ibuprofen use or acetaminophen use during the postpartum period. Standard blood pressure monitoring in the postpartum period will be followed to help determine if there is a significant rise in the women who use NSAIDS in the postpartum period versus those that use acetaminophen.

Groups will be divided into women with chronic hypertension, women with chronic hypertension with superimposed preeclampsia, women with preeclampsia without severe features, women with preeclampsia with severe features, women with gestational hypertension without severe range blood pressures, and women with gestational hypertension with severe range blood pressures.

Recruitment will last 36 months. Patients will be monitored during their postpartum stay (typical 2 days) with blood pressure measurements. An additional 12 months will be needed for data analysis and publication.

ELIGIBILITY:
Inclusion Criteria:

* vaginal delivery
* diagnosis of chronic hypertension, chronic hypertension with superimposed preeclampsia
* preeclampsia without severe features
* preeclampsia with severe features gestational hypertension without severe range blood pressures
* gestational hypertension with severe range blood pressures
* singleton pregnancies

Exclusion Criteria:

* Cesarean Delivery
* no diagnosis of hypertensive disorder
* chronic or acute renal disease
* allergy to ibuprofen or acetaminophen
* lupus
* multiple order pregnancies (twins, triplets)
* Narcotic addiction/ in treatment for substance abuse/ current prescription drug user/ current use of illegal drugs

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-10-08 (Actual); Study Completion 2017-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Goldkamp, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetaminophen: Women receiving acetaminophen for primary pain control following vaginal delivery.
- NSAID: Women receiving Ibuprofen for primary pain control following vaginal delivery.
Period: Overall Study
Arm/Group | Acetaminophen | NSAID
Started | 16 | 20
Completed | 16 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | NSAID | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Continuous [Mean (Full Range); unit: years] | 28 [16 to 44] | 25 [18 to 35] | 27 [16 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 20 | 36
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in the Mean Systolic Blood Pressure From Postpartum Day 1 Versus Postpartum Day 2.
Description: To determine if NSAIDS in the postpartum period raise blood pressure in women with a hypertensive disorder. The mean increase and standard deviation of each group (acetaminophen and NSAID/Ibupforen) was calculated when compairing systolic blood pressures from the first postpartum day to the second postpartum day. Day 1 is the mean of systolic blood pressures from 0 hours to 23 hours after delivery, and Day 2 is the mean of systolic blood pressures from 24 hours to 47 hours after delivery.
Time Frame: 2 days
Population: Mean difference day 1 compared to day 2 of systolic blood pressure
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Acetaminophen: Patients will be monitored for change in blood pressure
  Acetaminophen: Blood pressure will be monitored during postpartum stay (typical 2 days)
- NSAID: Patients will be monitored during their postpartum stay (typical 2 days) and then again at 1 week
  NSAID: Blood pressure will be monitored during postpartum stay (typical 2 days)
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 16 | 20
mmHg | 7.5 (13.8) | 5 (6.1)
Statistical Analysis 1: Comparison: Acetaminophen vs NSAID; Test type: Non-Inferiority; p < 0.05, Wilcoxon (Mann-Whitney); Mean Difference (Net) = 0.85

2. Secondary Outcome: Change in the Mean Diastolic Blood Pressure From Postpartum Day 1 Versus Postpartum Day 2.
Description: To determine if NSAIDS in the postpartum period raise blood pressure in women with a hypertensive disorder. The mean increase and standard deviation of each group (acetaminophen and NSAID/Ibupforen) was calculated when compairing diastolic blood pressures from the first postpartum day to the second postpartum day. Day 1 is the mean of diastolic blood pressures from 0 hours to 23 hours after delivery, and Day 2 is the mean of diastolic blood pressures from 24 hours to 47 hours after delivery.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- NSAID: Patients will be monitored during their postpartum stay (typical 2 days)
  NSAID: Blood pressure will be monitored during postpartum stay (typical 2 days)
Arm/Group | Acetaminophen | NSAID
Number analyzed (Participants) | 16 | 20
mmHg | 0.4 (11.1) | 2.7 (7.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Acetaminophen | NSAID
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20
Other Adverse Events (participants affected / at risk) | 0/16 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT02902172/Prot_SAP_000.pdf